CLINICAL TRIAL: NCT04806334
Title: Radiogenomics of Muscle Invasive Bladder Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Charles Rosser, Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IIT2020-22-Rosser
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer Stage II
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Not studying the MRI device; it is looking at feasibility of creating a radiogenomic workflow to learn about the correlation structure between the radiomic and genomic parameters of interest. The study is not an ACT but should be registered to meet ICMJE recommendations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 4D MRI of pelvis/bladder with genomic analysis of bladder tumor (Experimental): Patients with sessile appearing bladder masses who are destined to undergo transurethral resection of the bladder tumor (TURBT) and are felt by the treating physician to harbor MIBC will be enrolled. Prior to TURBT, ALL subjects will undergo axial imaging for clinical staging in the form of contrast enhanced MRI of the abdomen and pelvis (standard of care). The pelvic MRI will be multiparametric (mp)-4D MRI incorporating high resolution diffusion weighted imaging (HR-DWI). Both the abdominal and pelvic MRI will have an official interpretation by a radiologist, thus both can be used in the care of the subject. Next, ALL subjects will undergo TURBT at which time, voided urine, blood and fresh frozen bladder tumor will be collected. Follow-up pathology will be collected.
  Interventions: Diagnostic Test: MRI imaging of the pelvis/bladder; Diagnostic Test: genomic analysis of tumor

INTERVENTIONS:
Diagnostic Test: MRI imaging of the pelvis/bladder — The pelvic MRI will be multiparametric (mp)-4D MRI incorporating high resolution diffusion weighted imaging (HR-DWI).
Diagnostic Test: genomic analysis of tumor — Single cell RNA sequencing of transurethral resection of bladder tumor (TURBT)

SUMMARY:
Patients with suspected bladder tumor will undergo novel 4D MRI imaging along with single cell RNA sequencing in hopes of identifying a radiogenomic signature that can improve our staging of patients with muscle invasive bladder cancer.

DETAILED DESCRIPTION:
The study will accrue patients with sessile appearing bladder masses who are destined to undergo transurethral resection of the bladder tumor (TURBT) and are felt by the treating physician to harbor MIBC. Prior to TURBT, ALL subjects will undergo axial imaging for clinical staging in the form of contrast enhanced MRI of the abdomen and pelvis (standard of care). The pelvic MRI will be multiparametric (mp)-4D MRI incorporating high resolution diffusion weighted imaging (HR-DWI). Both the abdominal and pelvic MRI will have an official intrepretation by a radiologist, thus both can be used in the care of the subject. Next, ALL subjects will undergo TURBT at which time fresh frozen bladder tumor will be collected and subjected to single cell RNA sequencing. Pathologic stage will be determined and reported on both the TURBT specimen and radical cystectomy specimen. From the above radiogenomic data, the investigators will show feasibility, which the investigators will define as know-how to create a radiogenomic workflow and to learn about the correlation structure between the radiomic and genomic parameters of interest, which will allow the investigators to design future studies with adequate power.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be > 18 years of age.
2. Patient must have a sessile mass noted within the bladder on cystoscopy or imaging worrisome for bladder cancer, specifically MIBC.
3. Patient must agree to undergo staging which will include mp-4D MRI HR-DWI of the pelvis in addition to standard axial imaging of the abdomen.
4. Patient must be agreeable to undergo planned TURBT as part of the normal treatment course.
5. Patients must not have known or suspected primary urothelial carcinoma of the ureter, urethra, or renal pelvis.
6. Patients must not have known distant metastatic disease (e.g. pulmonary or hepatic metastases). Subjects with malignant lymphadenopathy in the abdomen or pelvis considered appropriate for radical cystectomy and lymphadenectomy with the goal of complete resection of all malignant disease are allowed.
7. Patients must not have had prior definitive treatment for bladder cancer.
8. Patients must not have clinically significant active infection or uncontrolled medical condition that would preclude participation in study.
9. Patients must not have any active malignancy other than urothelial carcinoma of the bladder that, in the opinion of the treating investigator, which could interfere with protocol treatment.
10. Patient must have adequate renal function: Serum creatinine < 2 mg/dL OR calculated CrCl > 30ml/min.
11. Patients must not have allergy or contraindication for MRI contrast/contrast dye.
12. Patients must not be under treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to TURBT.
13. Patient must not be adverse to undergo radical cystectomy as part of the normal treatment course if found to have MIBC.
14. Patients must have the ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

1. Persons with allergy to animal dander or animal-instigated asthma.
2. Patient must not have undergone a bladder biopsy or limited (incomplete) TURBT within 3 weeks (21 days) of the MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Rosser, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4D MRI of Pelvis/Bladder With Genomic Analysis of Bladder Tumor
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 4D MRI of Pelvis/Bladder With Genomic Analysis of Bladder Tumor
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 65.4545 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Proceed With MRI Imaging and Sequencing of Bladder Tumor
Description: Number of participants who proceed with radiogenomics analysis with useable data, that is a preliminary signature related to MIBC.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | 4D MRI of Pelvis/Bladder With Genomic Analysis of Bladder Tumor
Number analyzed (Participants) | 11
Participants | 10

ADVERSE EVENTS:
Time Frame: 84 weeks (study duration)
Arm/Group | 4D MRI of Pelvis/Bladder With Genomic Analysis of Bladder Tumor
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT04806334/Prot_SAP_000.pdf